CLINICAL TRIAL: NCT06705036
Title: Differential Study of Invasive Pituitary Adenomas in the Sellar and Cavernous Sinus Regions
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024683
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pituitary Tumor
Keywords: cavernous sinus; intrasellar
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Paired pituitary tumors from the sella and cavernous sinus of the same patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pituitary tumors in cavernous sinus group: The 20 pituitary tumor samples in this group were obtained from the cavernous sinus region removed during surgery and were paired with pituitary tumors in the intralellar region
  Interventions: Other: surgery
- pituitary tumors in sellar group: The 20 pituitary tumors in this group were obtained from intrasellar samples removed during surgery and were paired with pituitary tumors in the cavernous sinus region
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — Samples were obtained from patients by surgical excision and matched into groups

SUMMARY:
This study involves collecting paired tumor samples from intrasellar and cavernous sinus regions of 20 invasive pituitary tumor patients, preserving them at -80°C for quality multi-omics analysis. Proteomics and transcriptomics are employed to identify molecular differences, while imaging data (MRI/CT) assesses tumor morphology and invasion. In vitro experiments and mechanistic studies validate key findings, exploring how regional molecular differences affect tumor behavior. Data integration combines multi-omics and imaging features to uncover biomarkers and pathways associated with invasiveness and regional specificity, with statistical analysis ensuring significance and reliability.

DETAILED DESCRIPTION:
This study focuses on investigating the molecular and biological differences between the intrasellar and cavernous sinus regions in invasive pituitary tumors to uncover mechanisms driving their aggressiveness and to identify potential therapeutic targets.

The research begins with sample collection, selecting 20 patients with invasive pituitary tumors based on inclusion and exclusion criteria. Paired tumor tissue samples are collected from the intrasellar and cavernous sinus regions of each patient, ensuring accuracy and completeness. These samples are then preserved at -80°C to maintain quality for subsequent multi-omics analyses.

Next, multi-omics analysis is conducted to examine molecular differences. Proteomics, using technologies like mass spectrometry or protein arrays, identifies differentially expressed proteins between the two regions and assesses their biological functions. Transcriptomics, through RNA sequencing, explores significant differences in gene expression and associated pathways. These approaches aim to uncover molecular mechanisms driving the tumor's invasive behavior.

Imaging analysis complements the molecular studies by utilizing preoperative imaging data, such as MRI or CT, to evaluate tumor morphology, invasion depth, and the impact on surrounding tissues. This provides a structural and functional context for the molecular findings.

Biological experiments follow to validate key discoveries. In vitro studies using cell lines or organoid models test the role of specific genes or pathways identified in the omics analyses, such as through gene knockout or overexpression. Mechanistic studies focus on understanding how molecular differences between the intrasellar and cavernous sinus regions influence tumor behaviors like invasion, proliferation, and migration. Validation experiments, including Western blotting or immunofluorescence, confirm the expression patterns and regional specificity of significant molecules.

Finally, data integration and analysis combine findings from proteomics, transcriptomics, and metabolomics with imaging features. Bioinformatics tools integrate these datasets to identify biomarkers and pathways associated with the tumor's invasiveness and regional specificity. Imaging-omics integration links molecular profiles with imaging characteristics, while rigorous statistical analysis ensures the robustness and significance of the results, accounting for potential confounding factors.

This comprehensive approach aims to provide new insights into the biological mechanisms of invasive pituitary tumors and identify effective targets for innovative therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive pituitary tumors involving the cavernous sinus
2. Retrospective inclusion of patients who have signed informed consent forms for the donation of biological samples and health-related information
3. Age range: 18-80 years
4. Subjects are willing to participate in this study

Exclusion Criteria:

1. Non-invasive pituitary tumors
2. Pregnant or breastfeeding
3. Other conditions deemed unsuitable for participation in this clinical trial as assessed by the physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years who are clinically diagnosed with invasive pituitary tumors involving the cavernous sinus, have signed the informed consent form, and are willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in pathological features of tumors | 2025/12/01-2026/12/01
  Cell morphology, proliferation index (e.g. Ki-67), angiogenesis, and other pathological features of tumor tissue in different regions were analyzed to explore region-specific invasive manifestations

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No